CLINICAL TRIAL: NCT03304145
Title: Shared Decision Making in Pain Management Planning in Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carevive Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: G414
Record Dates: First submitted 2017-09-18; First posted 2017-10-06 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Cancer
Keywords: Treatment Care Planning
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The Carevive CPS — The Carevive Care Planning System (CPS) was developed to overcome challenges by providing an efficient, clinically integrated solution for both psychosocial and physical symptom distress screening and management through the delivery of personalized and evidence-based care plans at the point of care. The Carevive CPS simultaneously collects and aggregates discrete data for quality reporting and improvement.

SUMMARY:
The goal of this project is to evaluate the effectiveness of shared-decision-making (SDM) to manage chronic and breakthrough pain in patients with cancer. Providers will receive evidence-based education on shared decision-making strategies and comprehensive pain management at study start up. In addition, the information will be available on the Carevive platform for reference at the point of care. This multisite study will enroll 105 patients from three cancer institutions. This project will explore the SDM model using a touchscreen-based expanded pain assessment (EPA) to evaluate the impact of the shared-decision-making model on pain management, and explore its relationship to pain management care planning. Patients will use the Carevive Systems software in the clinic to answer questions regarding decision making preferences and complete a comprehensive assessment of their pain status. Treatment recommendations and a care plan will be provided to the patient at the time of the visit. At each clinic visit over 4 months, the patient will again complete the pain assessment and receive appropriate treatment recommendations and a revised care plan.

DETAILED DESCRIPTION:
Cancer-related pain is a significant clinical challenge that impacts patient outcomes and remains a significant problem for patients with cancer and their providers. The overall prevalence of cancer pain is high; a recent meta-analysis of 52 studies reported cancer pain prevalence ranging between 52%-77%. Another update reports rates of 39% after curative treatment, 55% during treatment, and 66% in advanced, metastatic or terminal disease. Moderate to severe pain was reported by 38% of all patients. Cancer pain may be cancer related, due to tumor burden causing bone, nerve, and/or organ compression, and/or treatment related, due to procedures, surgery, and side effects of chemotherapy or radiation. The prevalence of pain after breast cancer treatment ranges from 13%-93%; women with metastatic breast cancer often have bone pain from metastases and bisphosphonates. In a nationwide lung cancer study (N = 450), pain was reported by 92% of patients with advanced (stage IIIB/IV) NSCLC. Similar reports indicate pain ranges from 74% to 92%. Uncontrolled pain is the most common chief complaint of unplanned hospitalizations and readmissions. One study reported over half of the chief complaints provided by breast cancer patients with an emergency department (ED) visit were related to poorly controlled pain, respiratory or gastrointestinal symptoms. Finally, there is evidence that high symptom burden and poor management of symptoms and side effects also leads to suboptimal adherence to therapy.

Management of cancer pain requires that the patient be screened for the presence of pain at every clinical contact. A comprehensive assessment should be conducted if the patient is experiencing pain, including specific questions about location, duration, severity, quality, timing, duration, and impact on quality of life. A thorough understanding of pain also considers the temporal characteristics of the pain experience, determining if the pain is intermittent, that is bursts of severe pain without persistent chronic pain, persistent, with moderate to severe pain present throughout the day, and/or breakthrough pain described as the transient exacerbation of pain despite adequately controlled persistent pain. Breakthrough pain is reported to occur daily in 21%-70% of patients.

The prevalence of psychosocial and physical symptom distress in cancer is so compelling that the Commission on Cancer, the Oncology Nursing Society (ONS), American Society of Clinical Oncology (ASCO), and the National Committee for Quality Assurance (NCQA)'s Patient-Centered Oncology Care Standards all require distress screening that includes pain screening and assessment as a quality mandate in their accreditation and quality certification programs. In addition, the Centers for Medicare and Medicaid Services (CMMS)'s Oncology Care Model (OCM) requires a care management plan that includes symptom management. Included as quality measures are NQF384, pain intensity quantified, and NQF 383, plan of care for pain. In addition, value based care payment models seek to decrease emergency department (ED) visits and hospitalization days.

Carevive recently completed a project designed to improve adherence to quality metrics in breast cancer through education plus use of a tablet-based technology to screen for and manage identified distress, pain, and other breast cancer quality indicators available within ASCO's Quality Oncology Practice Initiative (QOPI) program. The Breast National Quality Standards project used QOPI metrics to evaluate outcomes of a CME intervention and use of the Carevive CPS. Preliminary data from this project showed improvement in key areas. Provider adherence to quality metrics was measured in 151 non-metastatic BC patients, 77 of which served as historical controls with no CME/clinical intervention, and 74 received the intervention after their provider participated in certified continuing medical education (CME) activities designed to educate about evidence-based assessment, decision-making, and management strategies for BC patients. Preliminary analysis showed that the intervention improved provider adherence to four pain quality measures: a. pain assessed by second office visit, b) pain intensity quantified by second office visit, c) plan of care documented, and d) pain assessed on either of the two most recent office visits. This project will build on that work to incorporate a comprehensive assessment and a more multi-faceted intervention that engages the care team in a SDM process around cancer pain management.

Along with an imperative to formalize a pain management plan is the rising importance of incorporating shared-decision-making, the cornerstone of patient centered care, into all care decisions. When making treatment decisions, the provider must incorporate current literature, patients' current clinical status, and patient preferences. One challenge with measuring quality through electronic chart abstraction is the difficulty of identifying when patient preference has influenced treatment decisions. Little data currently exist on the level of patient engagement in decision-making for pain management and the perception of patients with MBC, LC, or AC of shared-decision-making in developing a pain management care plan. Dr. Jeannine Brant and colleagues have developed the Pain Care Quality Survey (PainCQ©). The PainCQs are two tools that measure the quality of nursing and interdisciplinary care related to pain management as perceived by hospitalized individuals. These tools will be modified in this project to capture the variable contributions of different members in the care team, including oncology nursing staff.

Strategies to better manage chronic and breakthrough cancer pain are critical. Many cancer centers have incorporated distress screening using either the National Comprehensive Cancer Network (NCCN) Distress Thermometer or the Edmonton Symptom Assessment Scale (ESAS) tools. However, structured processes are typically lacking within the clinical workflow to seamlessly integrate and conduct a more in-depth assessment of those patients who score positively for pain. Processes and technologies that facilitate better integration of pain assessment and pain management care strategies into the oncology team's clinical workflow, while simultaneously integrating algorithms for treatment of pain have the potential to further drive evidence-based care.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be 18 years of age or older.
* Patient participants must have a diagnosis of cancer
* Patients must have screened positive for pain per a previous clinical assessment
* All participants must be able to understand English.

Exclusion Criteria:

* Any patient who cannot understand written or spoken English.
* Any prisoner and/or other vulnerable persons as defined by NIH (45 CFR 46, Subpart B, C and D).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Effect of pain care plan on pain outcomes | Year 1
  Pain intensity over time will be measured by the Sum of Pain Intensity Differences (SPID).

SECONDARY OUTCOMES:
Contribution of shared-decision-making on pain outcomes will be evaluated using the PainCQ© surveys | Year 1
  The PainCQ measures the patient's perception of the quality of pain management by the interdisciplinary team and whether the patient felt included in decision making.
Feasibility of the proposed shared decision-making model to effectively manage chronic pain experienced by patients with cancer | Year 1
  Participating OCM practices will complete a single feasibility assessment measuring completeness of each intervention tool

CONTACTS AND LOCATIONS:
Locations (1):
- Billings Clinic, Billings, Montana, United States

IPD SHARING:
Plan to Share IPD: No